CLINICAL TRIAL: NCT05283343
Title: Clinical Study of the Topcon Pachymeter TRK-3 to Evaluate Agreement and Precision
Status: Completed | Type: Observational
Sponsor: Topcon Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: THQ-2021-05
Record Dates: First submitted 2022-03-01; First posted 2022-03-16 (Actual); Last update posted 2022-07-22 (Actual); Status verified 2022-07

CONDITIONS: Corneal Thickness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Adults 20 years old or older
  Interventions: Device: SP-1P

INTERVENTIONS:
Device: SP-1P — A subject undergoes corneal thickness measurement with pachymeter.

SUMMARY:
Agreement and Precision of corneal thickness measurement (pachymetry) function of the test device TRK-3 and the predicate device SP-1P will be evaluated in volunteers, and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals who gave written informed consent to participate in the clinical trial by their free will.
2. Individuals who aged 20 years or older at the time of informed consent
3. Individuals who were deemed eligible for the study by the investigator for screening prior to enrollment.
4. Subjects who are able to comply with compliance items during participation in the clinical trial, undergo medical examination and examination specified in the protocol, and report subjective symptoms, etc.

Exclusion Criteria:

1. Individuals with ocular diseases that may affect corneal thickness measurement (blindness, corneal perforation, bullous keratopathy, nystagmus, etc.) or who have a history of ocular diseases and are considered by the investigator to be ineligible for participation in the study.
2. Individuals who have or are suspected of suffering from ocular or systemic infections.
3. Other persons who are judged by the investigator to be unfavorable candidates for the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects undergoing pachymetry measurement
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2021-11-27 (Actual); Primary Completion 2021-11-27 (Actual); Study Completion 2021-11-27 (Actual)

PRIMARY OUTCOMES:
Corneal thickness | 1 day
  Corneal thickness

CONTACTS AND LOCATIONS:
Locations (1):
- Samoncho Clinic, Tokyo, Japan